CLINICAL TRIAL: NCT04202601
Title: Efficacy and Safety Evaluation of Sintilimab in Combination With IBI310 as Treatment in Patients With Gastric Cancer
Brief Title: Efficacy and Safety Evaluation of Sintilimab in Combination With IBI310 as Treatment in Patients With EBV-Positive Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, MD,Professor,Chief of Department of GI Oncology,Peking University Cancer Hospital, Peking University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI310Y101
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Advanced Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neoadjuvant therapy group (Experimental)
  Interventions: Drug: Sintilimab; Drug: IBI310
- first-line therapy group (Experimental)
  Interventions: Drug: Sintilimab; Drug: IBI310
- ≥second-line therapy group (Experimental)
  Interventions: Drug: Sintilimab; Drug: IBI310

INTERVENTIONS:
Drug: Sintilimab — Arms 1: Neoadjuvant therapy group 20 patients Drug: Sintilimab Weight<60Kg: 3mg/kg Q3W Weight>=60Kg:200 mg Q3W on Day 1 by IV infusion; Intervention：Perioperative Sintilimab+IBI310 are administered for 1-3 (6-18 weeks) cycles followed by 4 postoperative cycles (12 weeks) with Sintilimab monotherapy .
  Arms 2: first-line therapy group, 30 patients Drug: Sintilimab Weight<60Kg: 3mg/kg Q3W Weight>=60Kg:200 mg Q3W on Day 1 by IV infusion; Intervention：Sintilimab + IBI310 are administered for 1-3 (6-18 weeks) cycles followed by Sintilimab monotherapy for up to 2 years.
  Arms 3: ≥second-line therapy group, 30 patients Drug: Sintilimab Weight<60Kg: 3mg/kg Q3W Weight>=60Kg:200 mg Q3W on Day 1 by IV infusion; Intervention：Sintilimab + IBI310 are administered for 1-3 (6-18 weeks) cycles followed by Sintilimab monotherapy for up to 2 years.
Drug: IBI310 — Arms 1: Neoadjuvant therapy group, 20 patients Drug: IBI310 1 mg/kg Q6W on Day 1 by IV infusion. Intervention：Perioperative Sintilimab+ IBI310 are administered for 1-3 (6-18 weeks) cycles followed by 4 postoperative cycles (12 weeks) with Sintilimab monotherapy .
  Arms 2: first-line therapy group, 30 patients Drug: IBI310 1 mg/kg Q6W on Day 1 by IV infusion. Intervention：Sintilimab + IBI310 are administered for 1-3 (6-18 weeks) cycles followed by Sintilimab monotherapy for up to 2 years.
  Arms 3: ≥second-line therapy group, 30 patients Drug: IBI310 1 mg/kg Q6W on Day 1 by IV infusion. Intervention：Sintilimab + IBI310 are administered for 1-3 (6-18 weeks) cycles followed by Sintilimab monotherapy for up to 2 years.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sintilimab+ IBI310 for EBV-Positive advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of unresectable locally advanced,recurrent or metastatic gastric or GEJ malignant tumor (including squamous carcinoma, adenocarcinoma, Signet-ring cell carcinoma).
* Confirmed EBV positive determined by in situ hybridization (ISH), analyzed with tumor tissue sample, either from a previous surgery or biopsy , within last 6 months
* Male or Female at least 18 years of age
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has adequate organ function.
* Expected survival>=12 weeks
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test at the timing of enrollment.
* Participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 6 months after the last dose of study medication.

Applied to Arms 1: Has histologically confirmed gastric/GEJ malignant tumor, and were regarded as having clinical stage T3-T4aN0M0 or T2～4aN+M0

Applied to Arms 2: Had no prior systemic treatment for metastatic disease.

Applied to Arms 3: Received ≥1 prior systemic treatment for metastatic disease.

Exclusion Criteria:

* Has received prior therapy with an anti-programmed death (PD)-1, antiPD-L1, anti-PD L2, anti-CTLA-4 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Is currently participating in and receiving study therapy ,except those in the survival follow up period of an investigational agent study or non-interventional study .
* Received systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 4 weeks of first dose. Inhaled or topical steroids ,adrenal replacement steroid doses and steroid of prevention allergic reaction of i.v. contrast agent are permitted in the absence of active autoimmune disease.
* Received a live vaccine within 4 weeks of the first dose of study medication or plan to receive live vaccine during study period.
* Has had major surgery (craniotomy, thoracotomy or laparotomy) within 4 weeks prior to first dose of study medication, or anticipation of the need for major surgery during the course of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-13 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Arms 1: Neoadjuvant therapy group | Approximately 40 months after the first participant is randomized
  Pathological complete regression (pCR):
  Pathological complete regression (pCR) is defined as the proportion of patients with pathological complete regression (TRG1a) over the total number of patients evaluated centrally by the study pathologist
Arms 2: first-line therapy group | Approximately 40 months after the first participant is randomized
  Objective response rate(ORR):
  Objective response rate(ORR) of Sintilimab in combination with IBI310 in all participants in this group.
Arms 3:≥second-line therapy group | Approximately 40 months after the first participant is randomized
  Objective response rate(ORR):
  Objective response rate(ORR) of Sintilimab in combination with IBI310 in all participants in this group.

SECONDARY OUTCOMES:
Arms 1: Neoadjuvant therapy group | Approximately 40 months after the first participant is randomized
  R0 resection rate
Arms 1: Neoadjuvant therapy group | Approximately 40 months after the first participant is randomized
  Event free survival(EFS)
Arms 1: Neoadjuvant therapy group | Approximately 40 months after the first participant is randomized
  Objective response rate(ORR)
Arms 1: Neoadjuvant therapy group | Approximately 40 months after the first participant is randomized
  Disease control rate(DCR)
Arms 1: Neoadjuvant therapy group | Approximately 40 months after the first participant is randomized
  Overall survival(OS)
Arms 1: Neoadjuvant therapy group | Approximately 40 months after the first participant is randomized
  Number of participants experiencing clinical and laboratory adverse events (AEs).
Arms 2: first-line therapy group | Approximately 40 months after the first participant is randomized
  Progression-free survival (PFS）
Arms 2: first-line therapy group | Approximately 40 months after the first participant is randomized
  Disease control rate (DCR）
Arms 2: first-line therapy group | Approximately 40 months after the first participant is randomized
  Overall survival (OS）
Arms 2: first-line therapy group | Approximately 40 months after the first participant is randomized
  ( Number of participants experiencing clinical and laboratory adverse events (AEs).
Arms 3:≥second-line therapy group | Approximately 40 months after the first participant is randomized
  Progression-free survival (PFS）
Arms 3:≥second-line therapy group | Approximately 40 months after the first participant is randomized
  Disease control rate (DCR)
Arms 3:≥second-line therapy group | Approximately 40 months after the first participant is randomized
  Overall survival (OS）
Arms 3:≥second-line therapy group | Approximately 40 months after the first participant is randomized
  Number of participants experiencing clinical and laboratory adverse events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No